CLINICAL TRIAL: NCT04649073
Title: A Multicenter, Uncontrolled, Nonrandomized, Open-Label, Phase 1/2 Trial Investigating the Safety and Efficacy of OPC 415 in MMG49 Antigen-Positive Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Safety and Efficacy Study of OPC-415 in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 415-102-00001
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OPC-415 (up to 1×10^7cells/kg) (Experimental)
  Interventions: Biological: OPC-415

INTERVENTIONS:
Biological: OPC-415 — OPC-415 (up to 1×10^7cells/kg) On 2 days

SUMMARY:
The purpose of this study is to evaluate the tolerability,safety and efficacy of OPC-415 in patients with relapsed and/or refractory Multiple Myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 80 (75 for the phase 1 part) years, both inclusive, at the time of consent
* Patients with a definitive diagnosis of active multiple myeloma
* Patients who have had 2 or more prior regimens (including all proteasome inhibitors, immunomodulators, and anti-CD38 antibody)
* Patients with relapsed and/or refractory Multiple Myeloma
* Patients who are positive for MMG49 antigen
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1. Those with an ECOG-PS score of 2 due solely to MM bone lesions can be enrolled
* Patients who are expected to survive for at least 3 months

Exclusion Criteria:

* Patients who are scheduled to receive high-dose chemotherapy in combination with autologous stem cell transplantation as the next treatment.
* Patients who have other active double/multiple cancers
* Patients on continuous and systemic (oral or intravenous) medication with corticosteroids or other immunosuppressive agents
* Patients with graft-versus-host disease that requires treatment.
* Patients who underwent a highly invasive and extensive surgical procedure within 2 weeks.
* Patients who previously underwent allogeneic stem cell transplantation or organ transplantation.
* Patients who underwent autologous stem cell transplantation within 90 days.
* Patients with systemic amyloidosis (except localized amyloidosis without organ derangement) or plasma cell leukemia.
* Patients with prior or current central nerve involvement in MM.
* Patients whose best ever response to MM treatment is PD.
* Patients who previously received gene therapy or cell therapy (except hematopoietic stem cell transplantation).
* Pregnant women, nursing mothers, or women with a positive pregnancy test.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2041-01 (Estimated)

PRIMARY OUTCOMES:
Phase1: Dose Limiting Toxicity | Day1~Day28
Phase2: Response rate | Day1~Day366
  The proportion of subjects who achieved partial response or better outcomes by central assessment based on IMWG Uniform Response Criteria for Multiple Myeloma will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Tokai University Hospital, Isehara-shi
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organization Okayama Medical Center, Okayama
  - Sapporo Medical University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya-ku
  - Osaka University Hospital, Suita-shi
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No
:The focus of this study is a rare disease.